CLINICAL TRIAL: NCT05961982
Title: Endoscopic Ultrasound-Guided Radiofrequency Ablation of Pancreatic Cysts - A Safety and Efficacy Trial (ERASE Study)
Brief Title: Evaluation of Endoscopic Ultrasound-Guided Radiofrequency Ablation for the Management of Pancreatic Tumors, ERASE Study
Acronym: ERASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Somashekar Krishna, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-22277; NCI-2023-04688 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT05916846 (obsolete NCT alias)
Record Dates: First submitted 2023-07-11; First posted 2023-07-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (EUS-RFA) (Experimental): Patients undergo standard of care EUS-FNA followed by EUS-RFA on study and may undergo repeat EUS-RFA or EUS-guided chemoablation during surveillance. Patients undergo MRI/MRCP, CT, or EUS-FNA at baseline and at follow-up timepoints.
  Interventions: Procedure: Chemical Ablation; Procedure: Computed Tomography; Other: Electronic Health Record Review; Procedure: Endoscopic Ultrasound-Guided Fine-Needle Aspiration; Procedure: Endoscopic Ultrasound-Guided Radiofrequency Ablation; Procedure: Magnetic Resonance Cholangiopancreatography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Chemical Ablation — Undergo EUS-guided chemoablation
  Other Names: ABLATION, CHEMICAL
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Procedure: Endoscopic Ultrasound-Guided Fine-Needle Aspiration — Undergo EUS-FNA
  Other Names: endoscopic ultrasound-guided fine needle aspiration; EUS-FNA
Procedure: Endoscopic Ultrasound-Guided Radiofrequency Ablation — Undergo EUS-RFA
  Other Names: EUS-RFA
Procedure: Magnetic Resonance Cholangiopancreatography — Undergo MRI/MRCP
  Other Names: MRCP
Procedure: Magnetic Resonance Imaging — Undergo MRI/MRCP
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This clinical trial evaluates the safety and effectiveness of endoscopic ultrasound-guided radiofrequency ablation (EUS-RFA) for the management of patients with pancreatic tumors (including cysts) performed during recommended surveillance endoscopic ultrasound examinations. Pancreatic tumors (cysts) can progress to pancreatic cancer at rate of more than 25% per year risk. Pancreatic cancer is a fatal disease that is difficult to diagnose at an early stage, and the five-year survival rate is currently less than 10%. It is projected to be the second leading cause of cancer-related mortality by the year 2030. A procedure known as radiofrequency ablation may help. Radiofrequency ablation is an established way to treat benign and cancerous tumors in the human body. In the last 5 years, radiofrequency ablation has been applied to treat precancerous tumors (including cysts) in the pancreas. This procedure implements a medical technology that destroys tumors in a much less invasive way compared to traditional surgical removal. By delivering a high-frequency alternating current, radiofrequency ablation uses electrical energy and heat to destroy cancer cells. Radiofrequency ablation is being recognized as a management option in patients with high-risk pancreatic tumors (cysts) but are not deemed surgical candidates. While surgical removal offers a chance of cure, pancreatic surgeries have 20-40% morbidity rate (short and long-term complication) and a 1-2% mortality rate in patients who are surgical candidates. Furthermore, radiofrequency ablation can potentially decrease the need for frequent imaging/surveillance of the pancreatic tumor (cyst). In patients with immediate prohibitive, but reversible risks for surgery, radiofrequency ablation of a high-risk tumors (cysts) can potentially prevent further progression of the lesion and bridge the time before the need for surgical resection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy of EUS-RFA of pancreatic cystic neoplasms (PCNs).

SECONDARY OBJECTIVES:

I. To assess the safety of EUS-guided RFA of PCNs. II. To assess the long-term response to EUS-RFA.

OUTLINE:

Patients undergo standard of care EUS-fine-needle aspiration (FNA) followed by EUS-RFA on study and may undergo repeat EUS-RFA or EUS-guided chemoablation during surveillance. Patients undergo magnetic resonance imaging (MRI)/magnetic resonance cholangiopancreatography (MRCP), computed tomography (CT), or EUS-FNA at baseline and at follow-up timepoints.

After completion of study treatment, patients are followed up every 3-6 months for cysts >= 3 cm or every 6-12 months for cysts < 3 cm for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* A diagnosis of a PCN confirmed by EUS-FNA including cyst fluid next generation sequencing (NGS) and/or EUS-guided needle-based confocal laser endomicroscopy (nCLE) and/or EUS- guided through-the-needle biopsy (TTNB)
* The pancreatic cystic lesion (PCL) measures at least 2 cm in diameter on either CT or MRI/MRCP or EUS and demonstrates concerning worrisome and/or high-risk features as defined by International Consensus Guidelines (2017 revised Fukuoka Guidelines)
* The patient is not a surgical candidate. Common clinical scenarios include -

  * Cirrhosis of the liver (common clinical scenario)
  * Advanced ( >= 75 years) age (common clinical scenario)
  * Morbid obesity
  * Significant cardiorespiratory comorbidity
  * Patient's choice (patient elects for non-surgical management)
  * Other significant comorbid conditions that impose prohibitive surgical risks
* Estimated life expectancy of at least 1 year
* Capable of giving written informed consent or has a legally authorized representative (LAR) to consent for them
* Women of childbearing potential must have a negative pregnancy test (serum/urine) on the day of treatment. Pregnancy testing is the routine standard of care practice in the endoscopy laboratory for all patients undergoing endoscopy and sedation for endoscopy
* The patient prefers non-surgical management after consultation with hepato-pancreato-biliary (HPB) surgery
* The patient is not a surgical candidate and has had prior attempts at ablation of the PCN by EUS-guided injection of chemotherapy (Ohio State University [OSU] Institutional Review Board [IRB] protocol 2020C0198)

Exclusion Criteria:

* A diagnosis of a benign or non-neoplastic PCL such as a pseudocyst confirmed by EUS-FNA including cyst fluid NGS and/or EUS-nCLE and/or EUS-TTNB
* A diagnosis of a malignant PCN confirmed by evidence of adenocarcinoma and/or invasive carcinoma and/or distant metastases
* Cysts or neuroendocrine tumors (NETS) involving or in close proximity to blood vessels, the biliary tree, or the main pancreatic duct where the zone of ablation is likely to compromise these structures
* Acute pancreatitis in the preceding 4 weeks prior to date of EUS-RFA
* Any evidence of severe or uncontrolled systemic diseases or laboratory finding that in the view of the investigator makes it unsafe for the patient to participate in the study
* Any psychiatric disorder making reliable informed consent impossible
* Pregnancy or breast-feeding
* Eastern Cooperative Oncology Group (ECOG) performance status 4
* Contraindication to general anesthesia after review by OSU Preoperative Assessment Clinic (OPAC)
* Cardiac implantable electrical devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of endoscopic ultrasound-guided radiofrequency ablation (EUS-RFA) | At 1 years after EUS-RFA
  Defined as at least a 50% decrease in the cyst diameter. Other markers of response to EUS-RFA will be evaluated by cross-sectional imaging and EUS: change in the diameter, morphology of cyst - fibrosis, septations, loculations, wall thickness, intracystic or mural nodules; cyst fluid aspiration (biopsy if there is fibrosis): next generation sequencing (NGS) - persistence or absence of mutations (molecular markers), cytology - results can include either: mucin, atypical/suspicious cells, necrotic material, or inflammatory debris, experimental: flow cytometry for immunological markers of antineoplastic response; serological changes: chromogranin A (for cystic-neuroendocrine tumor), and serum cancer antigen (CA) 19-9 (if elevated prior to intervention).

SECONDARY OUTCOMES:
Long-term response to EUS-RFA | At 2 and 3 years after EUS-RFA
  Defined as at least a 50% decrease in the cyst diameter. Durable response: Continued response with further decrease in cyst diameter beyond the first calendar year. The response will be evaluated by cross-sectional imaging and EUS: change in the diameter, morphology of cyst - fibrosis, septations, loculations, wall thickness, intracystic or mural nodules; cyst fluid aspiration (biopsy if there is fibrosis): NGS - persistence or absence of mutations (molecular markers), cytology - results can include either: mucin, atypical/suspicious cells, necrotic material, or inflammatory debris, experimental: flow cytometry for immunological markers of antineoplastic response; serological changes: chromogranin A (for cystic-neuroendocrine tumor), and serum CA 19-9 (if elevated prior to intervention).
Safety of EUS-guided RFA of pancreatic cystic neoplasms post procedure | Post-procedure (after EUS-RFA)
  Documented using the adverse events in gastrointestinal endoscopy classification for adverse events in gastrointestinal advanced endoscopy. Only grade II or higher degree of complications will be documented since patients are electively admitted after EUS-RFA for overnight observation. If patient has post-procedure acute pancreatitis, document severity based on Revised Atlanta Classification.
Safety of EUS-guided RFA of pancreatic cystic neoplasms at one year | at one year after EUS-RFA
  Documented using the adverse events in gastrointestinal endoscopy classification for adverse events in gastrointestinal advanced endoscopy. Only grade II or higher degree of complications will be documented since patients are electively admitted after EUS-RFA for overnight observation. If patient has post-procedure acute pancreatitis, document severity based on Revised Atlanta Classification.

CONTACTS AND LOCATIONS:
Overall Officials: Somashekar G Krishna, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu